CLINICAL TRIAL: NCT02963467
Title: Acute Effect of Smoking Cigarettes on Ventilation-Perfusion Ratio: A Pilot Study in Healthy Volunteers
Brief Title: Effect of Smoking on Ventilation-Perfusion Ratio
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ass.-Prof. Dr. Stefan Boehme, Assistent Professor, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1133/2013
Record Dates: First submitted 2016-11-04; First posted 2016-11-15 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Lung Disease
Keywords: multiple inert gas elimination technique; smoking; pulmonary disorder
MeSH Terms: conditions — Lung Diseases; Smoking | interventions — Tobacco Products; Smoking Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Volunteers - non-smokers (Other): control group: After baseline measurements V/Q will be measured by MIGET. After a 2 hour wash out period, the Volunteers will smoke a dummy cigarette. Then V/Q will be measured again after 15 minutes.
  Interventions: Procedure: "dummy cigarette"
- Healthy Volunteers - occasional smokers (Other): intervention: After baseline measurements V/Q will be measured by MIGET. After a 2 hour wash out period, the Volunteers will smoke 4 conventional cigarettes. Thereafter, V/Q will be measured again after 15, 30, 45, 60 and 120 minutes.
  Interventions: Procedure: cigarette
- Healthy Volunteers - heavy-smokers (Other): intervention: After baseline measurements V/Q will be measured by MIGET. After a 2 hour wash out period, the Volunteers will smoke 4 conventional cigarettes. Thereafter, V/Q will be measured again after 15, 30, 45, 60 and 120 minutes.
  Interventions: Procedure: cigarette

INTERVENTIONS:
Procedure: cigarette — smoking 4 conventional cigarettes
  Other Names: smoking
  Arms: Healthy Volunteers - heavy-smokers; Healthy Volunteers - occasional smokers
Procedure: "dummy cigarette" — smoking a "dummy cigarette"
  Other Names: smoking
  Arms: Healthy Volunteers - non-smokers

SUMMARY:
Smoking is one of the world's leading health hazards. Besides being a major risk factor in the etiology of COPD and lung cancer, cigarette smoke is also a causative agent lung diseases characterized by bronchiolar and interstitial inflammation. However, the associated lung pathology of smoking is not only a risk in the development of lung diseases, but also widely recognized as a major risk factor associated with perioperative respiratory and cardiovascular complications. Apart from the long term effects of cigarette smoke, acute effects of the inhalation of cigarettes smoke may influence the course of lung pathology. The inhalation of smoke causes inflammation in the lung by inducing chemotaxis and activation of neutrophils and macrophages and induces oxidative stress. As the acute inflammatory response to smoke inhalation seems to be the underlying mechanism for chronic diseases of smokers, exploring the field of the acute pulmonary changes after exposure to cigarette smoke is highly relevant. One reason for acute hypoxia and injury during smoking might be a severe mismatch of ventilation and perfusion of the lung. Using the multiple inert gas elimination technique (MIGET), a distribution of ventilation-perfusion ratios in the lung can be calculated by analyzing data on the retention and excretion of six infused inert gases. A saline solution containing the gases is infused intravenously. When passing through the lung the gases are either eliminated from the blood or retained depending on their partition coefficient and local V/Q ratio. The concentrations of the gases are measured in the mixed venous blood or the mixed expired gas and the arterial blood allowing for the calculation of retention and excretion and the derivation of V/Q distribution. MIGET is the experimental gold standard to determine the Ventilation-Perfusion ratio of the lung. The aim of this study is to show the acute effect of smoking on ventilation/perfusion ratio distribution in the lung in otherwise healthy smokers.

ELIGIBILITY:
Inclusion Criteria:

* normal body mass index (BMI)

Exclusion Criteria:

* Medical history of pulmonary or cardiovascular disease
* Family history of malignant hyperthermia, neuro-muscular disorders
* Known hypersensitivity to any of the inert gases or substances administered
* History of post operative nausea and vomiting
* Pregnancy (pregnancy test will be performed on study day)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
ventilation-perfusion ratio by MMIMS-MIGET | within a time-frame of 6 hours
  V/Q-ratio as well as shunt, low V/Q, normal V/Q and high V/Q i.e. deadspace will be assessed by micropore-membrane inlet mass-spectrometry multiple inert gas elimination technique (MMIMS-MIGET)

SECONDARY OUTCOMES:
serum nicotine by blood sampling | within a time-frame of 6 hours
  the serum nicotine level will be assessed by clinical chemistry

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No